CLINICAL TRIAL: NCT04851951
Title: Clinical Results Of Platelet Rich Plasma (PRP) One-Shot Injection For Supraspinatus Tendinosis, Our Experience At Short-Term Follow Up
Brief Title: Platelet Rich Plasma (PRP) One-Shot Injection For Supraspinatus Tendinosis
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other)
Responsible Party: Sponsor
Other Study IDs: PRP-shoulder
Record Dates: First submitted 2021-04-15; First posted 2021-04-21 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-04

CONDITIONS: Supraspinatus Tendinitis
Keywords: Supraspinatus tendinosis; PRP; Shoulder;

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients treated by one-shot PRP injection
  Interventions: Procedure: one-shot PRP injection

INTERVENTIONS:
Procedure: one-shot PRP injection — A single injection of PRP (7% concentrate) ml 4 was made in the Supraspinatus tendon and in the Subacromial space under ultrasound guidance.

SUMMARY:
It was conducted a prospective study with a series of 50 patients treated with PRP one-shot injection in patient affected by Supraspinatus Tendinosis. One independent observer performed clinical and functional evaluations at T0 (recruitment), T1 (one month after the injection), T2 (three months after the last injection) and T3 (six months after the last injection).

Constant Score, The Disabilites of the Arm,Shoulder and Hand Score (DASH) And Visual Analogue Scale (VAS) were administered at each evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old;
* Supraspinatus tendinosis detected by MRI.

Exclusion Criteria:

* Supraspinatus rupture;
* Previous shoulder surgery;
* Rotator cuff tears secondary to fracture;
* Hemoglobin <7 g/dL or Platelets < 30,000 microL;
* Active infection;
* Pregnant patients;
* Patients with hematologic and oncologic diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fifty (50) patients referring to the Orthopaedic and Trauma Unit of the local University Hospital between January 2018 and July 2020 with Supraspinatus tendinosis were prospectively recruited.
Sampling Method: Probability Sample
Enrollment: 48 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-07-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analogic Scale | Day 0; Month 1; Month 3; Month 6 (after the injection)
  The shoulder pain was quantified using the Visual Analogic Scale ranging from 0 (no pain) to 10 (worst imaginable pain).

CONTACTS AND LOCATIONS:
Locations (1):
- AOUC Policlinico di Bari - UOC Ortopedia e Traumatologia, Bari, Italy